CLINICAL TRIAL: NCT02667678
Title: 5 Years Follow-up Evaluation of Deterioration Kidney Biomarkers of HIV Patients : HIVOL 2 Study.
Brief Title: 5 Years Follow-up Evaluation of Deterioration Kidney Biomarkers of HIV Patients
Acronym: HIVOL2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1508032; 2015-001455-68 (EudraCT Number)
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: HIV
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort HIVOL, patients infected by HIV (Experimental): Patients enrolled in HIVOL cohort (study performed between 2011 and 2013) will be contacted to participate to HIVOL-2. The intervention will be blood and urinary samples, with the use of iohexol (Omnipaque®) to have an idea on renal plasmatic clearance.
  Interventions: Biological: Cohort HIVOL, patients infected by HIV

INTERVENTIONS:
Biological: Cohort HIVOL, patients infected by HIV — Researchers will take blood and urinary samples from the patients of the HIVOL cohort, to look at the renal clearance. The aim of this study is to check the renal function of the patients infected by HIV.
  Other Names: Blood and urinary samples

SUMMARY:
The aim of this study is to compare the biomarkers levels as IL-18, KIM-1 and Cystatin C for patients infected by HIV with failure in renal function at year 5. The main criterion will be a degradation of the glomerular filtration throughput measured. It will be compared to clinical scores of degradation risks of renal function for patients infected with HIV.

DETAILED DESCRIPTION:
The aim of this study is to compare the biomarkers levels as IL-18, KIM-1 and Cystatin C for patients infected by HIV with failure in renal function at year 5. The main criterion will be a degradation of the glomerular filtration throughput measured. It will be compared to clinical scores of degradation risks of renal function for patients infected with HIV.

From 2011 to 2013, researchers realized a study called HIVOL, on the diagnostic performance of GFR (Glomerular Filtration Rate) estimators in patients infected with HIV. It lead to a publication in AIDS, retaken in the rational of recommendations of Infectious Diseases Society of America for the Chronic Renal Diseases support for patients infected with HIV.

235 patients were involved, for everyone researchers have a GFR measure (by Iohexol plasmatic clearance) and urinary and plasma samples.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated or entitled to a social security scheme
* Patient HIV infected
* Patient included in the HIVOL cohort with a GFR measure available
* Patients who have given their consent in writing

Exclusion Criteria:

* Pregnant or lactating women
* Patients treated with metformin
* Patients with a known allergy, regardless the type of allergy
* Patients with a history of thyroid dysfunction
* Any biological anomaly in the selection, which in the opinion of the investigator, may indicate a contraindication to the patient's participation in this study
* Degradation recent (not older than three months) of renal function defined as the degradation of more than 25 % GFR.
* Estimated GFR of less than 15 mL / min / 1.73m2
* History of major immediate or delayed skin reaction known to the injection of iodinated contrast medium (OMNIPAQUE®)
* Manifest thyrotoxicosis
* Hypersensitivity to the active substance or to any of the excipients (OMNIPAQUE®)
* Patient who expressed his refusal to participate in the study
* Patient justice under protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Stage of chronic kidney disease (according to the Glomerular Filtration Rate) | Day 1
  The aim of this study is to compare the level of biological biomarkers as microalbuminuria, proteinuria, KIM-1, IL-18, and Cystatin C with the level of this markers 5 years ago, for the HIVOL study performed between 2011 and 2013. These levels will allow the researchers to have an idea concerning the renal function of the patients followed.

CONTACTS AND LOCATIONS:
Overall Officials: GAGNEUX-BRUNON Amandine, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No